CLINICAL TRIAL: NCT02507856
Title: Prospective Record Of the Use of Dabigatran in Patients With Acute Stroke or TIA
Acronym: PRODAST
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hans Diener, Prof. Dr. med., University Hospital, Essen
Other Study IDs: PRODAST
Record Dates: First submitted 2015-07-16; First posted 2015-07-24 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Brain Ischemia With Non-valvular Atrial Fibrillation; Transient Ischemic Attack With Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- investigational group: early/late dabigatran
- control group: vitamin k antagonist (vka)

SUMMARY:
The multi-center, prospective PRODAST study is investigating patients with non-valvular atrial fibrillation (AF) who experienced an ischemic stroke or a transient ischemic attack (TIA) recently (≤ 1 week) both with and without previous oral anticoagulation. It consists of a baseline visit and a 3 months central follow-up for patients who were discharged with dabigatran, vitamin K-antagonists, antiplatelets only, or no oral antithrombotic treatment at all. Thus, data on the use of dabigatran and vitamin K-antagonists in routine clinical practice will be collected to describe how dabigatran is prescribed and used in the population of AF patients with recent cerebrovascular events and how these factors influence important outcome and safety events. The utilization of dabigatran will be assessed with regards to treatment persistence, compliance, proportion of patients discontinuing treatment and reason for discontinuation as well clinical endpoints such as major bleeding, stroke or systemic embolism. Due to the fact that patients will be treated according to local medical practice it is possible that medication will be changed during the observation period. In the follow-up, data from the first as well as from the second prescribed medication will be used in the study. To explore a long-term effect of anticoagulation, survival up to one year will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at enrollment
* Male or female patient willing and able to provide written informed consent for data transmission. For patients who are not legally competent to sign this informed consent for data transmission exceptions/special cases are described in the protocol.
* Patient with ischemic stroke or TIA within the last 7 days.
* Patient diagnosed with non-valvular AF. Documentation of AF by 12 lead ECG, ECG rhythm strip, monitor print-out, pacemaker/ICD electrocardiogram, Holter ECG (duration of AF episode at least 30 seconds) or written physician´s diagnosis prior to index event needed for all enrolled patients.

Exclusion Criteria:

* Presence of any mechanical heart valve, or valve disease that is expected to require valve replacement intervention (surgical or non-surgical) during the next 3 months.
* Current participation in any randomized clinical trial of an experimental drug or device.
* Women of childbearing age without anamnestic exclusion of pregnancy or not using an effective contraception or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent (≤ 1 week from index) ischemic stroke or TIA and with confirmed non-valvular AF (documented by 12 lead ECG, ECG rhythm strip, pacemaker/ICD electrocardiogram, or Holter ECG) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 10044 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Major bleeding event rate | from study inclusion up to 3 months
  Major bleeding event rate within 3 months following the index event (= stroke or TIA)

SECONDARY OUTCOMES:
Complications during hospitalisation | from index event up to 1 week
  Complications during hospitalisation before study inclusion (= signature of informed consent)
Number of participants with newly occurring or recurrent strokes | from study inclusion up to 3 months
  Stroke (hemorrhagic, ischemic or uncertain classification)
Severity of stroke assessed by modified Rankin Scale (mRS) | from study inclusion up to 3 months
Number of participants with newly occurring or recurrent TIA | from study inclusion up to 3 months
  transient ischemic attack
Number of participants with systemic embolism | from study inclusion up to 3 months
Number of participants with pulmonary embolism | from study inclusion up to 3 months
Number of participants with myocardial infarction | from study inclusion up to 3 months
Life-threatening bleeding events | from study inclusion up to 3 months
Any cause of death | from study inclusion up to 3 months
  any cause of death (non-vascular, vascular or unknown cause)
Point in time for withdrawal/change of medication | from study inclusion up to 3 months
Reason for withdrawal/change of medication | from study inclusion up to 3 months
Patient compliance | from study inclusion up to 3 months
Treatment persistence | from study inclusion up to 3 months
(Serious) Adverse Events (AE/SAE) | from study inclusion up to 3 months
Survival one year after study inclusion | up to 1 year from study inclusion
  any cause of death (non-vascular, vascular or unknown cause)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Diener, Prof. Dr., Study Director — University Hospital, Essen
Locations (90):
- Germany (90):
  - Klinikum Altenburger Land GmbH, Altenburg
  - Kreisklinik Altötting, Altötting
  - Schön Klinik Bad Aibling, Bad Aibling
  - Hochtaunus-Kliniken gGmbH, Krankenhaus Bad Homburg, Bad Homburg
  - Neurologische Klinik Bad Neustadt a. d. Saale, Bad Neustadt an der Saale
  - Klinikum Bayreuth, Bayreuth
  - Vivantes Auguste-Viktoria Klinikum, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Vivantes Humboldt Klinikum GmbH, Berlin
  - Evangelisches Krankenhaus Bielefeld gGmbH, Bielefeld
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil GmbH, Bochum
  - St. Josef Hospital Ruhr University Bochum, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Knappschaftskrankenhaus Bottrop GmbH, Bottrop
  - Klinikum Bremerhaven-Reinkenheide gGmbH, Bremerhaven
  - Krankenhaus Buchholz und Winsen gGmbH, Buchholz
  - Evangelisches Krankenhaus Castrop-Rauxel, Castrop-Rauxel
  - Allgemeines Krankenhaus Celle, Celle
  - REGIOMED-Kliniken - Klinikum Coburg, Coburg
  - Universitätsklinikum Köln, Cologne
  - Krankenhaus St. Elisabeth gGmbH, Damme
  - Klinikum Dortmund gGmbH, Dortmund
  - Städtisches Klinikum Dresden-Neustadt, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Evangelisches Klinikum Niederrhein gGmbH, Duisburg
  - Klinikum Emden, Hans-Susemihl Krankenhaus, Emden
  - Alfried Krupp Krankenhaus Rüttenscheid, Essen
  - University Hospital Essen, Department of Neurology, Essen
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fulda gAG, Fulda
  - Evangelische Kliniken Gelsenkirchen gGmbH, Gelsenkirchen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Klinikum Oberberg - Kreiskrankenhaus Gummersbach GmbH, Gummersbach
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - UKH Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Wandsbek, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Evangelisches Krankenhaus Hattingen gGmbH, Hattingen
  - Krankenhaus Agatharied GmbH, Hausham
  - Universitätsklinikum Heidelberg, Heidelberg
  - Evangelisches Krankenhaus Herne, Herne
  - BDH-Klinik Hessisch-Oldendorf GmbH, Hessisch Oldendorf
  - Klinikum Ibbenbüren GmbH, Ibbenbueren
  - Klinikum Idar-Oberstein GmbH, Idar-Oberstein
  - SHR Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Alexianer Krefeld GmbH, Krankenhaus Maria-Hilf, Krefeld
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Klinikum Main-Spessart, Krankenhaus Lohr, Lohr
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Sana Kliniken Luebeck GmbH, Lübeck
  - Städtisches Klinikum Lüneburg gGmbH, Lüneburg
  - St.-Marien-Hospital GmbH, Lünen
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum Merzig, Merzig
  - Mühlenkreiskliniken AöR, Johannes Wesling Klinikum Minden, Minden
  - St. Josef Krankenhaus GmbH Moers, Moers
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - UKM Universitätsklinikum Münster, Münster
  - Dietrich-Bonhoeffer-Klinikum Neubrandenburg, Neubrandenburg
  - Klinikum Osnabrück GmbH, Osnabrück
  - Klinikum Vest GmbH, Behandlungszentrum Knappschaftskrankenhaus Recklinghausen, Recklinghausen
  - Imland Klinik Rendsburg, Rendsburg
  - Klinikum Saarbrücken gGmbH, Saarbrücken
  - Nordwest-Krankenhaus Sanderbusch, Sande
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - ASKLEPIOS Kliniken Schildautal Seesen, Seesen
  - Kreisklinikum Siegen, Siegen
  - Medinos Kliniken Sonneberg, Sonneberg
  - Klinikum Stuttgart - Katharinenhospital, Stuttgart
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - Asklepios Fachklinikum Teupitz, Teupitz
  - Universitätsklinikum Tübingen, Tübingen
  - RKU - Universitäts- und Rehabilitationskliniken Ulm gGmbH, Ulm
  - Ammerland Klinik GmbH, Westerstede
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Sana HANSE-Klinikum Wismar, Wismar
  - Klinikum Wolfsburg, Wolfsburg
  - Rhein-Maas-Klinikum GmbH, Würselen
  - Universitätsklinikum Würzburg AöR, Würzburg

REFERENCES:
- [Derived] Grosse GM, Husing A, Stang A, Kuklik N, Brinkmann M, Grond M, Rollnik JD, Marquardt L, Kraft A, Schlemm E, Eggers C, Eschenfelder CC, Weimar C, Diener HC. Prior Anticoagulation and Risk of Hemorrhagic Transformation in Acute Stroke: A Post Hoc Analysis of the PRODAST Study. J Am Heart Assoc. 2025 Feb 4;14(3):e037014. doi: 10.1161/JAHA.124.037014. Epub 2025 Feb 3. PMID 39895532

DOCUMENTS (1):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02507856/Prot_001.pdf